CLINICAL TRIAL: NCT01719991
Title: Pragmatic Evaluation of Case Management and Self-management Support for Vulnerable People With Chronic Diseases in Primary Care
Brief Title: Vulnerable Patients in Primary Care: Nurse Case Management and Self-management Support
Acronym: V1SAGES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Agence de la Sante et des Services Sociaux du Saguenay-Lac-Saint-Jean (Other); Centre de santé et de services sociaux de Chicoutimi (Other); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Catherine Hudon, MD, Pr, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FRSQ-26758
Record Dates: First submitted 2012-10-25; First posted 2012-11-01 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Diseases
Keywords: Primary care; Self-management; Self-support; Nurse case management
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nurse case management and self-management support (Experimental): The first component of the intervention is the monitoring offered under the case management process. The second component of the intervention consists of group meetings (10-12 people) for self-management support in accordance with the stanford model. A sample of patients in each of the four FMGs (n = 126) will be recruited. These patients will receive the intervention for six months.
  Interventions: Other: Nurse case management and self-management support
- Control group (No Intervention): Patients in the control group (n = 121) will receive the usual care for six months and then the same intervention as the experimental group for the next five months (waiting list control group).

INTERVENTIONS:
Other: Nurse case management and self-management support — Case management: The intervention will focus on four main components: (1) A thorough evaluation of the patient's needs and resources; (2) Establishing and maintaining a patient-centered, individualized service plan (ISP); (3) Coordination of services among partners; and (4) Self-management support for patients and their families.
  Self-management support: A standardized six-week program with interactive weekly group meetings led by two volunteer peer helpers (appointed trainers), who themselves have a chronic disease.
  Arms: Nurse case management and self-management support

SUMMARY:
The purpose of this study is to implement a pragmatic intervention in four (4) family medicine groups(FMGs) in the region of Saguenay-Lac-Saint-Jean (Quebec, Canada)for patients with chronic diseases.

DETAILED DESCRIPTION:
Chronic diseases represent a major health burden worldwide. Some people with chronic diseases require a higher level of care due to personal characteristics that increase their vulnerability. For these patients, nurse effective case management in primary care are associated with positive outcomes. Moreover, self-management programs, such as the standford program developed by the School of Medicine at the University of Standford in California (USA), are also recognized for their benefits on patients with chronic diseases.

The aim of our project is to implement, within four (4) FMGs of the region of Saguenay-Lac-Saint-Jean , a practical intervention involving case management by a nurse to promote interdisciplinary person-centered monitoring and self-management support for highly vulnerable individuals with chronic diseases (diabetes, cardiovascular diseases, respiratory diseases, musculoskeletal diseases and/or chronic pain).

The objectives of our study : 1) To analyze the implementation of the intervention in the participating FMGs in order to determine how the various contexts have influenced the implementation and the observed effects; 2) To evaluate the proximal and intermediate effects of the intervention on patients; 3) To conduct an economic analysis of the effectiveness and cost-benefit of the intervention.

The analysis of the implementation will be conducted using realistic evaluation approaches and participatory practice within four categories of key players (FMG stakeholders, FMG/health center managers, patients and their families, health center partners or communities). The data will be obtained through individual or group interviews, literature reviews and documentation from the intervention undertaken. The evaluation of the effects in patients will be based on a pragmatic randomized experimental design before and after (six months) with delayed intervention in the control group. Economic analysis will include a cost-effectiveness analysis and a cost-benefit analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient of the participating FMGs
* Aged between 25 and 80 years
* Affected by chronic disease (diabetes, cardiovascular diseases, respiratory diseases, musculoskeletal diseases and/or chronic pain)
* Identified as a frequent user of health services (by a health care provider or/and a software)

Exclusion Criteria:

* Patient unable to provide consent
* With cognitive impairment
* With uncontrolled psychiatric illness
* Patient with a prognostic of less than one years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in patient perception of personal self-efficacy at 6 months | 6 months
  The patient capacity to self-management measured by the Self-Efficacy for Managing Chronic Disease instrument.
Change in patient perception of self-management practice at 6 months | 6 months
  The patient capacity to manage their condition and their physical and psychological reaction measured by a subscale of the Health Education Impact Questionnaire (HEIQ).
Change in patient perception of health behaviours at 6 months | 6 months
  Fruit and vegetable consumption, smoking status, alcohol consumption, healthy weight and physical activity.
Change in patient perception of activation at 6 month | 6 months
  Patient knowledge, skills and self-confidence in self-management measured by the Patient Activation instrument.
Change in patient perception of psychological distress at 6 months | 6 months
  Measured by the Psychological Distress instrument.

SECONDARY OUTCOMES:
Change in patient perception of empowerment at 6 months. | 6 months
  Health education impact measured by the Health Education Impact Questionnaire (HEIQ).
Change in patient perception of quality of life at 6 months | 6 months
  Measured by the 12-Item Short Form Health Survey
Change in use of health services at 6 months | 6 months
  Measured by hospitalizations, emergency room visits and health services use(e.g., psychosocial services or specialized services related to the specific chronic disease.

OTHER OUTCOMES:
Socioeconomic status | 2 weeks before the intervention
Health literacy status | 2 weeks before the intervention
  The degree to which individuals have the capacity to obtain, process and understand basic health information and services needed to make appropriate health decisions measured by the Newest Vital Sign.
Mental health status | 2 weeks before the intervention
  Measured by the Hospital Anxiety and Depression Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Hudon, PhD, Principal Investigator — Université de Sherbrooke; Maud-Christine Chouinard, PhD, Principal Investigator — Université du Québec à Chicoutimi
Locations (2):
- Canada (2):
  - Centre de santé et de services sociaux Lac-Saint-Jean-Est, Alma, Quebec
  - Centre de santé et de services sociaux de Chicoutimi, Chicoutim, Quebec

REFERENCES:
- [Derived] Hudon C, Chouinard MC, Dubois MF, Roberge P, Loignon C, Tchouaket E, Lambert M, Hudon E, Diadiou F, Bouliane D. Case Management in Primary Care for Frequent Users of Health Care Services: A Mixed Methods Study. Ann Fam Med. 2018 May;16(3):232-239. doi: 10.1370/afm.2233. PMID 29760027
- [Derived] Couture EM, Chouinard MC, Fortin M, Hudon C. The relationship between health literacy and patient activation among frequent users of healthcare services: a cross-sectional study. BMC Fam Pract. 2018 Mar 9;19(1):38. doi: 10.1186/s12875-018-0724-7. PMID 29523095
- [Derived] Couture EM, Chouinard MC, Fortin M, Hudon C. The relationship between health literacy and quality of life among frequent users of health care services: a cross-sectional study. Health Qual Life Outcomes. 2017 Jul 6;15(1):137. doi: 10.1186/s12955-017-0716-7. PMID 28683743
- [Derived] Chouinard MC, Hudon C, Dubois MF, Roberge P, Loignon C, Tchouaket E, Fortin M, Couture EM, Sasseville M. Case management and self-management support for frequent users with chronic disease in primary care: a pragmatic randomized controlled trial. BMC Health Serv Res. 2013 Feb 7;13:49. doi: 10.1186/1472-6963-13-49. PMID 23391214